CLINICAL TRIAL: NCT06170814
Title: Investigation of the Effects of Different Focuses of Attention on Functional Walking and Balance in Children With Cerebral Palsy
Brief Title: Effects of Different Focuses of Attention on Walking and Balance in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Gazi University
Other Study IDs: Cerebral palsy and gait
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Palsy; Gait, Hemiplegic; Balance
Keywords: cerebral palsy; External focus; internal focus; gait and balance
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- external odak: Exercise will be done for approximately 40 minutes, 3 days a week for 6 weeks. Ramps, obstacle jumping, stairs and tracks will be built to improve walking and balance functions. During exercises, attention is directed to movement and an environmental stimulus in the external focus of attention.
  Interventions: Other: Exercise
- internal focus: Exercise will be done for approximately 40 minutes, 3 days a week for 6 weeks. Ramps, obstacle jumping, stairs, and tracks will be built to improve walking and balance functions. In internal focus during exercises, attention is directed directly to body movements.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise will be done for approximately 40 minutes, 3 days a week for 6 weeks. Ramps, obstacle jumping, stairs and tracks will be built to improve walking and balance functions. One group will be given external focus stimuli, the other group will be given internal focus stimuli.

SUMMARY:
This study was planned to examine the effects of different focuses (external and internal focus)of attention on functional walking and balance in children with cerebral palsy. Individuals with CP between the ages of 6-18 will be included in the research. It was planned to include 24 individuals in total, 12 individuals in each group.

DETAILED DESCRIPTION:
In the external focus of attention (EF), attention is directed to movement and an environmental stimulus. In the internal focus (IF), attention is directed directly to body movements. In revealing positive effects in external focus; Methods such as metaphor, analogy, imaginary objects, mental analogies can be used. Adopting an External focus of attention (focusing on the effects of movements on the object or environment), as opposed to an Internal focus of attention (focusing on body movements), has been found to significantly improve performance on a variety of tasks. Walking and balance are essential for activities of daily living and social participation; Therefore, it is often considered one of the most important activities in daily life. Walking and balance is an automatic rhythmic motor behavior controlled mostly by subcortical brain regions. Automaticity means that walking can be performed without requiring attention. Although it seems like a very simple activity, it is actually a very complex chain of movements in which the brain, spinal cord, muscles, bones and joints work together in coordination. However, movement, balance and gait disorders cause individuals with CP to spend more energy, deteriorate their mobility and decrease their independence. Although the beneficial effects of EF have not yet been demonstrated for every population, the constrained action hypothesis encourages the use of an EF for teaching motor skills. Looking at the literature, the effects of EF on the development of motor performance in children with cerebral palsy have not been examined. Therefore, this study aims to examine the effects of external focus of attention on gait and balance.

Individuals with CP between the ages of 6-18 will be included in the research. After the purpose and scope of the study are explained to all individuals and their families who agree to participate in the study, their families will be asked to read and sign the volunteering form. All individuals who meet the inclusion criteria will be randomly divided into 2 groups (external focus and internal focus). It was planned to include 24 individuals in total, 12 individuals in each group. The same evaluations will be made to all individuals participating in the study by a physiotherapist who is an expert in the field. In addition to conventional physiotherapy for 6 weeks, individuals will be included in an exercise program that focuses on external and internal attention for 30 minutes a day, 3 days a week. Evaluation of walking function will be done with the C-Mill Walking Training System. Balance function will be performed by standing on one leg, pediatric berg balance scale and functional reaching tests.Independence Pediatric Functional Independence Scale will be evaluated with.Trunk control, trunk control measurement scale will be evaluated with.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with spastic type cerebral palsy between the ages of 6-18
* Volunteerism of the family and individuals to participate in the study
* Being at levels I and II according to the Gross Motor Classification System
* Having the cognitive development to be cooperative

Exclusion Criteria:

* Having undergone any orthopedic and/or neurological surgery in the last 6 months,
* Having hearing and/or vision loss that would prevent participation in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with hemiparatic cerebral palsy between the ages of 6 and 18 will be included in the study.
  In order to perceive the commands during the exercise, the children participating in the study must have a level of cognitive development to be cooperative.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Gait | 6 week
  Walking function will be evaluated twice with the C-Mill Walking Training System, before and at the end of treatment (6 weeks of treatment).

SECONDARY OUTCOMES:
balance | 6 week
  Balance function will be evaluated twice, before and at the end of treatment (6 weeks of treatment), with the one-leg standing test and the functional reaching test.
Trunk control measurement scale | 6 week
  trunk control, trunk control measurement scale will be evaluated with.
Pediatric Functional Independence Scale | 6 week
  Independence, Pediatric Functional Independence Scale will be evaluated with.
pediatric berg balance scale | 6 week
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabia ERASLAN, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beauchet O, Berrut G. [Gait and dual-task: definition, interest, and perspectives in the elderly]. Psychol Neuropsychiatr Vieil. 2006 Sep;4(3):215-25. French. PMID 16945851
- [Result] Yamada M, Raisbeck LD, Porter JM. The Effects of Using Imagery to Elicit an External Focus of Attention. Res Q Exerc Sport. 2021 Sep;92(3):559-565. doi: 10.1080/02701367.2020.1733455. Epub 2020 Mar 6. PMID 32142388
- [Result] Bunger A, Urfer-Maurer N, Grob A. Multimethod Assessment of Attention, Executive Functions, and Motor Skills in Children With and Without ADHD: Children's Performance and Parents' Perceptions. J Atten Disord. 2021 Feb;25(4):596-606. doi: 10.1177/1087054718824985. Epub 2019 Jan 30. PMID 30700232
- [Result] Blank R, Barnett AL, Cairney J, Green D, Kirby A, Polatajko H, Rosenblum S, Smits-Engelsman B, Sugden D, Wilson P, Vincon S. International clinical practice recommendations on the definition, diagnosis, assessment, intervention, and psychosocial aspects of developmental coordination disorder. Dev Med Child Neurol. 2019 Mar;61(3):242-285. doi: 10.1111/dmcn.14132. Epub 2019 Jan 22. PMID 30671947
- [Derived] Zorlular R, Akinci M, Elbasan B. Effects of focus of attention on gait parameters and balance performance in children with unilateral cerebral palsy: a randomized controlled trial. Disabil Rehabil. 2026 Feb;48(3):829-841. doi: 10.1080/09638288.2025.2548412. Epub 2025 Aug 21. PMID 40839080